CLINICAL TRIAL: NCT07052539
Title: The Epidemiology and Pathophysiology of Kidney Disease in HFpEF With Obesity
Status: Recruiting | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1040
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease; Heart Failure With Preserved Ejection Fraction (HFPEF); Obesity (Disorder)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (3):
- Healthy Participants
  Interventions: Other: High protein and sodium meal
- Obese Participants without HFpEF
  Interventions: Other: High protein and sodium meal
- HFpEF and Obese Participants
  Interventions: Other: High protein and sodium meal

INTERVENTIONS:
Other: High protein and sodium meal — Meal with 1g/kg protein content and 3900mg sodium

SUMMARY:
This research study wants to learn about Chronic Kidney Disease (CKD) with Obesity, and Heart Failure with preserved Ejection Fraction (HFpEF) and better ways to evaluate these diseases. HFpEF means that the heart is not able to fill properly with blood while it is resting so the amount of blood pumped out to the body is less than it would be if it was filling properly. The study is being done to describe the differences in how the kidneys handle protein and salt in participants with HFpEF and obesity compared to healthy persons.

ELIGIBILITY:
Criteria for Cohort 1: Healthy Participants

Inclusion Criteria:

* Adults 18-75 years old
* Normal kidney function
* No heart failure
* BMI 25-30kg/m2

Exclusion Criteria:

* Diagnosis of chronic illness
* eGFR<60mL/min/1.73m2
* Pregnancy or breast feeding
* History of cutaneous or allergic reaction to iodine-based products of contrast dyes
* Hemoglobin levels <7mg/dL
* Acute illness or hospitalization event within 3 months
* Unable to stop NSAIDs
* Comorbid conditions: MM, amyloidosis, pheochromocytoma, SCD, metastatic brain lesions, advanced kidney disease, liver dysfunction, endotoxemia, hyperthyroidism
* Current use of nicotine or recreational drugs, chronic drinker

Criteria for Cohort 2: Obese Participants without HFpEF

Inclusion Criteria:

* Adults 18-75 years old
* eGFR >= 60 mL/min/1.73m2
* BMI > 35 kg/m2

Exclusion Criteria:

* Diagnosis of Heart Failure
* Diagnosis of chronic illness
* eGFR<60mL/min/1.73m2
* Pregnancy or breast feeding
* History of cutaneous or allergic reaction to iodine-based products of contrast dyes
* Hemoglobin levels <7mg/dL
* Acute illness or hospitalization event within 3 months
* Unable to stop NSAIDs
* Comorbid conditions: MM, amyloidosis, pheochromocytoma, SCD, metastatic brain lesions, advanced kidney disease, liver dysfunction, endotoxemia, hyperthyroidism
* Current use of nicotine or recreational drugs, chronic drinker

Criteria for Cohort 3: HFpEF and Obese Participants

Inclusion Criteria:

* Adults 18-75 years old
* eGFR >= 60 mL/min/1.73m2
* BMI > 35 kg/m2
* Diagnosis of HFpEF (chart diagnosis, LVEF > 55% on echo, H2FPEF score 6-9 or HFA-PEFF score 5 or 6

Exclusion Criteria:

* NYHA class III/IV
* Urinary retention screen +
* Mobility issues
* History of RRT or kidney transplant
* Acute illness/hospitalization in the past 3 months
* History of cancer, chemo, or XRT
* Pregnant/breastfeeding
* History of allergies to contrast
* Hemoglobin < 7
* Comorbid conditions: MM, amyloidosis, pheochromocytoma, SCD, metastatic brain lesions, advanced kidney disease, liver dysfunction, endotoxemia, hyperthyroidism
* Unable to stop NSAIDs
* Current use of nicotine or recreational drugs, chronic drinker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling ambulatory participants who have HFpEF and obesity. We will compare with health participants and participants with obesity but without HFpEF.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in measured GFR | 5 hours
Change in urine sodium excretion | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marissa C Tio, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No